CLINICAL TRIAL: NCT00261664
Title: Empowering Elders Through Technology
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Collaborators: University of Pennsylvania (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 49150
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: telehomecare

SUMMARY:
Telehomecare is a technology that individuals use in their homes to communicate with health providers electronically. This technology can help them function at a higher level and avoid undesirable hospitalizations by making changes in their everyday behaviors, but research is needed to understand how telehomecare supports health behavior change and leads to improved health status.

The hypothesis being tested is that the use of an electronic method of monitoring and transmitting health information facilitates patient empowerment, with subsequent effects on the patient's ability to manage her/his treatment regimen more effectively. The study will explore the relationship between telehomecare and acquisition of knowledge, and will show whether changes in knowledge levels translate to changes in behaviors and improved health outcomes. The effects of two different telehomecare systems (nurse-directed vs. patient-directed) on knowledge, self-management, and health status will be compared. A further goal is to illuminate the attitudes of physicians regarding the use of telehomecare in the treatment of their elderly, community dwelling patients.

Results will inform managers and policymakers who are responsible for integrating eHealth mechanisms into chronic disease protocols, funding health care programs, and creating policies that support the use of information technology by all Americans.

DETAILED DESCRIPTION:
This study, funded by the Robert Wood Johnson Foundation through its Health e-Technologies Initiative (www.hetinitiative.org) is investigating the impact of telehomecare on health outcomes of persons with heart failure. The study began on September 1, 2003 and ends on February 28, 2006.

This study targets elderly persons with congestive heart failure (CHF), a major health problem affecting more than 4 million Americans. The research hypothesis being tested is that the use of an electronic method of monitoring and transmitting health information facilitates patient empowerment, with subsequent effects on the patient's ability to manage her/his treatment regimen more effectively. The study will explore the linkages between telehomecare and acquisition of knowledge, and will show whether changes in knowledge levels translate to changes in behaviors and improved health outcomes.

The effects of two different telehomecare systems (nurse-directed vs. patient-directed) on knowledge, self-management, and health status will be compared. A further goal is to illuminate the attitudes of physicians regarding the use of telehomecare in the treatment of their elderly, community dwelling patients.

Specific objectives are:

1. To evaluate the impact of telehomecare on patients' knowledge and self-management of heart failure, and cardiovascular health outcomes;
2. To compare the effect of two different telehomecare systems on patients' knowledge and self-management of heart failure, and cardiovascular health outcomes;
3. To investigate how the personal characteristics of older persons influence human-computer interaction and user satisfaction;
4. To describe and predict the attitudes and intentions of physicians regarding the use of telehomecare applications; and,
5. To analyze relationships among individual characteristics, information use, self-management of heart-failure and health status.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of congestive heart failure
* must have telephone line in home

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290
Dates: Start 2003-09; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Self-management of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Dansky, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States